CLINICAL TRIAL: NCT03352830
Title: Understanding Adoption of Clean Cookstoves
Brief Title: Encouraging LPG Adoption in Ghana: A Factorial Randomized Clinical Trial to Enhance LPG Adoption & Sustained Use
Acronym: ELAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Darby Jack, Assistant Professor of Environmental Health Sciences, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AAAO4965; R01ES024489 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-11-24 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Behavior, Consumer; Health Knowledge, Attitudes, Practice; Health Attitude
Keywords: household air pollution; health promotion; clean cookstove adoption; clean cookstove sustained use
MeSH Terms: conditions — Consumer Behavior; Behavior

STUDY DESIGN:
Masking Description: Masking is not feasible for this intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): All individuals in each arm will receive a new LPG cookstove. The control arm will receive an orientation for safe operation of the new LPG stove. Participants in the control arm will, however, receive no other intervention.
- No Delivery, Educational Intervention (Experimental): All individuals in each arm will receive a new LPG cookstove. This intervention arm receives a health promotion intervention based on the Risks, Attitudes, Norms, Ability, and Self-Regulation (RANAS) model.
  Interventions: Behavioral: RANAS Behavior Change Intervention
- Delivery, No Educational Intervention (Experimental): All individuals in each arm will receive a new LPG cookstove. This intervention arm receives free direct delivery of their LPG cylinder refills upon demand.
  Interventions: Other: Infrastructural Intervention - Direct Delivery
- Agent Delivery, Educational Intervention (Experimental): All individuals in each arm will receive a new LPG cookstove. This intervention arm receives free direct delivery of their LPG cylinder refills upon demand. Participants in this arm also receive a health promotion intervention based on the Risks, Attitudes, Norms, Ability, and Self-Regulation (RANAS) model.
  Interventions: Behavioral: RANAS Behavior Change Intervention; Other: Infrastructural Intervention - Direct Delivery

INTERVENTIONS:
Behavioral: RANAS Behavior Change Intervention — The Risks, Attitudes, Norms, Abilities, and Self-Regulation (RANAS) Model is a health behavior change intervention, which has been successfully used in the area of water, sanitation, and hygiene. It draws from numerous health behavior theories, including the Theory of Planned Behavior, the Health Action Process, and the Health Belief Model. The model posits that the five factor blocks (risks, attitudes, norms, abilities, and self-regulation) that must be aligned toward the new behavior in order to influence change. A series of activities target each block accordingly.
  Arms: Agent Delivery, Educational Intervention; No Delivery, Educational Intervention
Other: Infrastructural Intervention - Direct Delivery — Product demand is influenced, in part, by accessibility. Investigators are testing the degree to which this is true for liquefied petroleum gas (LPG) by establishing a direct delivery system for communities randomized to this treatment arm. Individuals in these communities are able to contact a 'delivery agent', contracted by the Kintampo Health Research Centre, who will: 1) retrieve their cylinder, 2) refill with LPG, and 3) return to the participant. The cost of delivery is free to the participant (paid by the study), but the participant is expected to fully pay for their own LPG.
  Arms: Agent Delivery, Educational Intervention; Delivery, No Educational Intervention

SUMMARY:
Household air pollution (HAP) is a top-priority public health problem in developing countries. According to the most recent comparative risk assessment, 3.5 million people die prematurely each year as a result of HAP exposures. While uncertainties remain regarding causal links between HAP exposures and health, the time is ripe for focused research into effective interventions. Limited past research has shown that the demand for clean cookstoves is low, and that households continue to use traditional hearths even when they have clean stoves. The investigators propose to harness an existing cohort in Ghana to study factors that increase the adoption of clean cookstoves, and to test strategies to promote adoption and continued use.

DETAILED DESCRIPTION:
Health conditions resulting from household air pollution (HAP) are responsible for approximately 3.9 million premature deaths each year. Exposure to HAP is the third largest preventable contributor to illness worldwide. Even so, HAP exposures persist since 3 billion individuals worldwide continue to rely on biomass fuel for cooking and heating, especially in the developing world. Though the transition away from traditional biomass stoves is projected curb the health effects of HAP by mitigating exposure, the benefits of newer clean cookstove technologies can only be fully realized if use of these stoves is exclusive and sustained. Most studies indicate that the provision of clean cookstoves to these individuals is, on its own, insufficient to encourage and foster adoption. In order to better understand how to promote clean cookstove adoption, the proposed study aims to (1) develop an educational intervention to promote clean cookstove adoption and sustained use and (2) determine the influence of liquid petroleum gasoline (LPG) accessibility on product demand.

Households enrolled into the control and the BioLite arms of GRAPHS (the parent study) will receive clean LPG cookstoves for their participation in the study (clinicaltrials.gov registration: NCT01335490). The objective of this study is to test the relative impact of two approaches to encourage stove use: providing a behavior change intervention and offering convenient access to LPG refueling. The investigators hypothesize that these interventions will increase overall use of LPG cook stoves.

Prior evidence on the role of health information in promoting the adoption of health-promoting technology is limited, and the results are mixed. Although little work has been done to investigate the importance of accessibility to sustained use of cookstoves, accessibility remains one of the basic market drivers of product demand.

A total of 27 communities will be cluster randomized, with 979 study households nested throughout the sites. The study arms will be arranged as a 2x2 factorial design, with approximately equal numbers of households in each arm.

ELIGIBILITY:
Inclusion criteria -- an individual is eligible to participate in the study if she:

* Previously participated in the Ghana Randomized Air Pollution and Health Study (GRAPHS; NCT01335490)
* Was originally randomized to the Biolite or Control arms of GRAPHS
* Currently resides in the Kintampo Health Research Centre study area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Minutes of LPG Use (via SUMS) | 10 months
  The investigators will measure stove use via iButton stove use monitors. The study period will be broken into two time spans, the first and second five months of the study. Our primary outcome of interest will be aggregated minutes of stove use over the second five months of the study.

SECONDARY OUTCOMES:
Amount of LPG refueled (via weight) | 10 months
  The investigators will measure stove use alternatively via biweekly weighing of LPG cylinders. The study period will be broken into two time spans, the first and second five months of the study. Our secondary outcome of interest will be aggregated kilograms of LPG over the second five months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Darby Jack, PhD, Principal Investigator — Columbia University
Locations (2):
- Columbia University Medical Center, New York, New York, United States
- Kintampo Medical Research Center, Kintampo, Ghana

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared between the study teams at the Kintampo Health Research Center and Columbia University. This data will not include medical or clinical information.
Supporting Information: SAP, CSR
Time Frame: The information will become available to the Columbia University team upon study completion.
Access Criteria: Data will be stripped of personally-identifiable information and encrypted before sharing.

REFERENCES:
- [Background] Smith KR, Bruce N, Balakrishnan K, Adair-Rohani H, Balmes J, Chafe Z, Dherani M, Hosgood HD, Mehta S, Pope D, Rehfuess E; HAP CRA Risk Expert Group. Millions dead: how do we know and what does it mean? Methods used in the comparative risk assessment of household air pollution. Annu Rev Public Health. 2014;35:185-206. doi: 10.1146/annurev-publhealth-032013-182356. PMID 24641558
- [Background] Bonjour S, Adair-Rohani H, Wolf J, Bruce NG, Mehta S, Pruss-Ustun A, Lahiff M, Rehfuess EA, Mishra V, Smith KR. Solid fuel use for household cooking: country and regional estimates for 1980-2010. Environ Health Perspect. 2013 Jul;121(7):784-90. doi: 10.1289/ehp.1205987. Epub 2013 May 3. PMID 23674502
- [Background] Lewis JJ, Bhojvaid V, Brooks N, Das I, Jeuland MA, Patange O, Pattanayak SK. Piloting improved cookstoves in India. J Health Commun. 2015;20 Suppl 1:28-42. doi: 10.1080/10810730.2014.994243. PMID 25839201
- [Background] Rehfuess E, Mehta S, Pruss-Ustun A. Assessing household solid fuel use: multiple implications for the Millennium Development Goals. Environ Health Perspect. 2006 Mar;114(3):373-8. doi: 10.1289/ehp.8603. PMID 16507460
- [Background] Jack DW, Asante KP, Wylie BJ, Chillrud SN, Whyatt RM, Ae-Ngibise KA, Quinn AK, Yawson AK, Boamah EA, Agyei O, Mujtaba M, Kaali S, Kinney P, Owusu-Agyei S. Ghana randomized air pollution and health study (GRAPHS): study protocol for a randomized controlled trial. Trials. 2015 Sep 22;16:420. doi: 10.1186/s13063-015-0930-8. PMID 26395578
- [Background] Mosler HJ. A systematic approach to behavior change interventions for the water and sanitation sector in developing countries: a conceptual model, a review, and a guideline. Int J Environ Health Res. 2012;22(5):431-49. doi: 10.1080/09603123.2011.650156. Epub 2012 Jan 31. PMID 22292899
- [Background] Lewis JJ, Pattanayak SK. Who adopts improved fuels and cookstoves? A systematic review. Environ Health Perspect. 2012 May;120(5):637-45. doi: 10.1289/ehp.1104194. Epub 2012 Feb 1. PMID 22296719
- [Derived] Carrion D, Dwommoh R, Tawiah T, Agyei O, Agbokey F, Twumasi M, Mujtaba M, Jack D, Asante KP. Enhancing LPG adoption in Ghana (ELAG): a factorial cluster-randomized controlled trial to Enhance LPG Adoption & Sustained use. BMC Public Health. 2018 Jun 4;18(1):689. doi: 10.1186/s12889-018-5622-3. PMID 29866127